CLINICAL TRIAL: NCT01395368
Title: Cognitive Speed as an Objective Measure of Tinnitus
Acronym: COMeT
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Jay F. Piccirillo, MD, Professor, Washington University School of Medicine, Washington University School of Medicine
Other Study IDs: 201103191
Record Dates: First submitted 2011-07-13; First posted 2011-07-15 (Estimated); Results first posted 2012-08-23 (Estimated); Last update posted 2012-08-23 (Estimated); Status verified 2012-07

CONDITIONS: Tinnitus
Keywords: subjective; unilateral; bilateral; non-pulsatile; 6 month's duration or longer
MeSH Terms: conditions — Tinnitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Brain Speed Test: Brain Speed Test

SUMMARY:
Tinnitus, commonly referred to as "ringing in the ears", affects 50 million people in the United States and is recognized as a major public health concern. Tinnitus is the most frequent cause of service-connected disability claims among war veterans. Tinnitus remains a subjectively diagnosed entity. There is no standardized objective method of diagnosing tinnitus or describing the functional impact of the condition. Currently, physicians have to rely on patient-based self reports. Without an objective method of diagnosing tinnitus and describing the functional implications, adequate treatment delivery is also hampered since there is no way to objectively stratify patients into severity groups and assess response to treatment. Because tinnitus is known to negatively affect cognition through the ventral attention networks and the prefrontal cortex, measuring cognitive processing speed is a possible way to objectively measure tinnitus. This study builds on previous work the investigators have done that utilized a quick, easily accessible measure of auditory processing speed. That earlier study showed a correlation between that measure and self reported measures of tinnitus severity, and this study attempts determine a more precise estimate of that correlation. It also better validates those results by including a traditional neurocognitive measuring cognitive speed and by controlling for the presence of depression and somatoform disorders.

DETAILED DESCRIPTION:
This was a cross-sectional study designed to investigate the relationship that self-reported tinnitus severity has with cognitive processing speed and psychiatric factors

ELIGIBILITY:
Inclusion Criteria:

* Participants must be between the ages of 18 and 80.
* Participants must have subjective, unilateral or bilateral, non-pulsatile tinnitus of 6 month's duration or longer.
* Participants must be able to read, write and speak using the English language.
* Participants must be able to read and follow the instructions for both computerized tests, "The Brain Speed Test" and "The 60 Second Brain Game."
* Participants must be able to provide written informed consent.

Exclusion Criteria:

* Participants with tinnitus related to Workman's Compensation Claim or other litigation-related situations.
* Participants with active diagnoses of any acute or chronic brain-related neurological conditions that alter normal brain anatomy or function including Parkinson's disease, Multiple Sclerosis, Alzheimer's Disease, cerebral infarcts, traumatic brain injury, history of brain tumor(s), epilepsy, or dementia.
* Participants with tinnitus related to retrocochlear lesions, cochlear implants, or other known anatomic/structural lesions of the brain, skull-base, temporal bone or ear.
* Participants who have a hearing threshold above 90 dB on any of the tested frequencies during audiometry.
* Participants unable to hear the highest volume of the computer-based objective assessments.
* Participants taking any medications that may affect or alter cognition including but not limited to sedatives, hypnotics, narcotics, or opiates.
* Participants with any medical condition the PI determines would compromise the safety of the participant or complicate the interpretation of the study results.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include men and women between the ages of 18-80 years who have subjective, unilateral or bilateral, non-pulsatile tinnitus of 6 month's duration or longer.
Sampling Method: Non-Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2011-06; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jay F Piccirillo, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University, St Louis, Missouri, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from Washington University's Volunteer for Health office, the audiology division and the otolaryngology faculty clinical practices at Washington University Department of Otolaryngology-Head and Neck Surgery, including the PI's population of tinnitus patients.
Groups:
- Tinnitus: Participants must be between the ages of 18 and 80. Participants must have subjective, unilateral or bilateral, non-pulsatile tinnitus of 6 month's duration or longer.
Period: Overall Study
Arm/Group | Tinnitus
Started | 108
Completed | 92
Not Completed | 16
Not completed — Physician Decision | 14
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Tinnitus
Number analyzed (Participants) | 92
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 83
  >=65 years | 9
Age Continuous [Mean (Standard Deviation); unit: years] | 53 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 63
Region of Enrollment [Number; unit: participants]
  United States | 92

OUTCOME MEASURES:

1. Primary Outcome: Brain Speed Test
Description: Standardized Z-scores of the Brain Speed Test (BST-Z scores) calculated based on age group-matched normal population data were used for analysis in order to control for the impact of age on test scores. Age-standardized Z-scores, which reflect the distance from the mean in standard deviation values, allow for the comparison of scores across age groups. A z-score of 0 indicates a value of the average, while absolute z-score values above 2 indicate observations significantly different from normal populations.
Time Frame: Participants completed brain speed test on the same day as enrollment. No follow-up required.
Population: Number of participants who completed the study with the exception of 4 subjects whose data was excluded due to the fact that they were younger than the the normative age-specific data available and BST Z-scores were not able to be calculated.
Measure: Mean (95% Confidence Interval); unit: z-score
Arm/Group | Tinnitus
Number analyzed (Participants) | 92
z-score | -0.09 [-0.23 to 0.05]

ADVERSE EVENTS:
Arm/Group | Tinnitus
Serious Adverse Events (participants affected / at risk) | 0/92
Other Adverse Events (participants affected / at risk) | 0/92

LIMITATIONS AND CAVEATS:
Tinnitus subjects with moderate or greater depression were excluded from the study. This study may not be reflective of the population of bothersome tinnitus patients due to this exclusion

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No